CLINICAL TRIAL: NCT01343485
Title: Staying on Track: Increasing Completion of the HPV Vaccine Series With the Use of an Innovative Patient and Provider Information and Tracking Tool
Brief Title: Innovative Tool to Increase Completion of Human Papillomavirus (HPV) Vaccine Series
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Planned Parenthood Federation of America (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Johanna Morfesis, Director of Research, Planned Parenthood Federation of America
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PPFA-Merck-38068
Record Dates: First submitted 2011-04-26; First posted 2011-04-28 (Estimated); Results first posted 2013-12-02 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-04

CONDITIONS: GARDASIL Vaccination
Keywords: Human papillomavirus (HPV) vaccine; Gardasil vaccine
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control, standard care for HPV vaccine (No Intervention): Study participants in control sites will receive standard care for HPV vaccine administration and follow-up per PPFA protocol
- Intervention, computer reminder system (Experimental): Study participants in the intervention sites will receive standard care for HPV vaccine administration per PPFA protocol, reminder messages for subsequent vaccination appointments, and real-time determination of financial assistance for HPV vaccine.
  Interventions: Behavioral: Computer reminder system

INTERVENTIONS:
Behavioral: Computer reminder system — Intervention sites will receive computer kiosk with study specific software to assist in reminding study participants to return for HPV vaccine series
  Arms: Intervention, computer reminder system

SUMMARY:
Planned Parenthood Federation of America's (PPFA) Medical Affairs Division will conduct a prospective, cluster randomized trial to determine which factors influence the acquisition of the second and third human papillomavirus (HPV) vaccine doses among young women ages 19 to 26. This descriptive and interventional study will provide data to assess impact of a computerized tool upon HPV vaccine series completion. The interventional aspect of this study includes determination of patient assistance and provider support programs applicable to each woman's situation as well as the implementation of a computer software system for customized patient reminders.

ELIGIBILITY:
Inclusion Criteria:

* Female;
* Age 19-26;
* Fluent in English;
* Seeking services for anything except pregnancy or abortion on the day of the visit
* No previous vaccinations for HPV
* No contraindication for HPV vaccine (includes a severe allergic reaction to yeast, amorphous aluminum hydroxyphosphate sulfate, and polysorbate 80.)
* Access to phone, text, mail, email, or facebook
* Not wanting to become pregnant in the next 8 months;
* Not planning on moving from the area in the next 8 months
* Willing to be contacted for follow-up over the next 8 months.

Exclusion Criteria:

* Women below 19 or above 26.
* Male
* Women who have one or more of HPV vaccination.
* Women who have a contraindication for HPV vaccine.
* Women who do not have access by phone, mail, email, Twitter or Facebook for follow up.
* Women who are not fluent in English
* Pregnant women or those intending on becoming pregnant during the study period.
* Women who will be moving from the area and unable to return for follow up over the course of the study (approximately 8 months).
* Severe mental impairment and unable to give Informed Consent.

Ages: 19 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 365 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashlesha Patel, MD, MPH, Principal Investigator — Planned Parenthood Federation of America, Inc.
Locations (9):
- United States (9):
  - Planned Parenthood of Arizona, Glendale, Arizona
  - Planned Parenthood of Rocky Mountains, Arvada, Colorado
  - Planned Parenthood of Rocky Mountains, Denver, Colorado
  - Family Planning Clinic of the John H. Stroger Jr. Hospital of Cook County, Chicago, Illinois
  - Planned Parenthood of Central North Carolina, Chapel Hill, North Carolina
  - Planned Parenthood of North Carolina, Charlotte, North Carolina
  - Planned Parenthood Association of Utah, Ogden, Utah
  - Planned Parenthood Association of Utah, South Jordan, Utah
  - Planned Parenthood of Greater Northwest, Seattle, Washington

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Recommended adult immunization schedule--United States, 2011. MMWR Morb Mortal Wkly Rep. 2011 Feb 4;60(4):1-4. No abstract available. PMID 21381442
- [Background] Chao C, Velicer C, Slezak JM, Jacobsen SJ. Correlates for completion of 3-dose regimen of HPV vaccine in female members of a managed care organization. Mayo Clin Proc. 2009 Oct;84(10):864-70. doi: 10.4065/84.10.864. PMID 19797775
- [Background] Dempsey A, Cohn L, Dalton V, Ruffin M. Patient and clinic factors associated with adolescent human papillomavirus vaccine utilization within a university-based health system. Vaccine. 2010 Jan 22;28(4):989-95. doi: 10.1016/j.vaccine.2009.10.133. Epub 2009 Nov 17. PMID 19925899
- [Background] Jain N, Euler GL, Shefer A, Lu P, Yankey D, Markowitz L. Human papillomavirus (HPV) awareness and vaccination initiation among women in the United States, National Immunization Survey-Adult 2007. Prev Med. 2009 May;48(5):426-31. doi: 10.1016/j.ypmed.2008.11.010. Epub 2008 Dec 6. PMID 19100762
- [Background] Neubrand TP, Breitkopf CR, Rupp R, Breitkopf D, Rosenthal SL. Factors associated with completion of the human papillomavirus vaccine series. Clin Pediatr (Phila). 2009 Nov;48(9):966-9. doi: 10.1177/0009922809337534. Epub 2009 May 29. No abstract available. PMID 19483128
- [Background] Orenstein WA, Mootrey GT, Pazol K, Hinman AR. Financing immunization of adults in the United States. Clin Pharmacol Ther. 2007 Dec;82(6):764-8. doi: 10.1038/sj.clpt.6100401. Epub 2007 Oct 31. PMID 17971821
- [Background] Sandfort JR, Pleasant A. Knowledge, attitudes, and informational behaviors of college students in regard to the human papillomavirus. J Am Coll Health. 2009 Sep-Oct;58(2):141-9. doi: 10.1080/07448480903221368. PMID 19892651
- [Derived] Patel A, Stern L, Unger Z, Debevec E, Roston A, Hanover R, Morfesis J. Staying on track: a cluster randomized controlled trial of automated reminders aimed at increasing human papillomavirus vaccine completion. Vaccine. 2014 May 1;32(21):2428-33. doi: 10.1016/j.vaccine.2014.02.095. Epub 2014 Mar 13. PMID 24631099
- See also: Planned Parenthood Federation of America — https://www.plannedparenthood.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention, Computer Reminder System: Study participants in the intervention sites will receive standard care for HPV vaccine administration per PPFA protocol, reminder messages for subsequent vaccination appointments, and real-time determination of financial assistance for HPV vaccine.
  Computer reminder system : Intervention sites will receive computer kiosk with study specific software to assist in reminding study participants to return for HPV vaccine series
Period: Overall Study
Arm/Group | Control, Standard Care for HPV Vaccine | Intervention, Computer Reminder System
Started | 185 | 180
Completed | 36 | 46
Not Completed | 149 | 134

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control, Standard Care for HPV Vaccine | Intervention, Computer Reminder System | Total
Number analyzed (Participants) | 185 | 180 | 365
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 185 | 180 | 365
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.64 (2.15) | 23.17 (2.18) | 23.41 (2.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 185 | 180 | 365
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 185 | 180 | 365

OUTCOME MEASURES:

1. Primary Outcome: On-time Completion of the Human Papillomavirus Vaccine Series
Time Frame: 32 weeks after receipt of initial vaccine
Measure: Number; unit: participants
Arm/Group | Control, Standard Care for HPV Vaccine | Intervention, Computer Reminder System
Number analyzed (Participants) | 185 | 180
participants | 36 | 31

ADVERSE EVENTS:
Arm/Group | Control, Standard Care for HPV Vaccine | Intervention, Computer Reminder System
Serious Adverse Events (participants affected / at risk) | 0/185 | 0/180
Other Adverse Events (participants affected / at risk) | 0/180 | 0/185

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No